CLINICAL TRIAL: NCT04823299
Title: AWARE-2 - Randomized Controlled Trial Ablation Strategy for Paroxysmal Atrial Fibrillation - Trigger and Substrate Guided Wide Area Radiofrequency Ablation Compared to Pulsed Field Ablation Pulmonary Vein Isolation
Brief Title: Randomized Controlled Trial- Ablation Strategy for Paroxysmal Atrial Fibrillation - Trigger and Substrate Guided Wide Area Radiofrequency Ablation Compared to Pulsed Field Ablation Pulmonary Vein Isolation
Acronym: AWARE-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: v21022021
Record Dates: First submitted 2021-03-23; First posted 2021-03-30 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation; Catheter Ablation; Radiofrequency Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Single-blind, prospective, randomized
Who Masked: Participant
Masking Description: Participant only blinded to the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoballoon ablation (Active Comparator): Cryoballoon Pulmonary Vein Isolation-Wide area circumferential ablation (WACA)
  Interventions: Procedure: Cryoballoon ablation
- RF based WACA ± EP testing guided ablation of non-PV triggers of AF and low voltage area ablation (Experimental): Radiofrequency wide area circumferential ablation (WACA) ± electrophysiological testing guided ablation of non-pulmonary vein triggers of AF and low voltage area ablation
  Interventions: Procedure: Radiofrequency catheter ablation +EPS guided trigger and substrate ablation

INTERVENTIONS:
Procedure: Cryoballoon ablation — Cryoballoon pulmonary vein isolation ablation
  Arms: Cryoballoon ablation
Procedure: Radiofrequency catheter ablation +EPS guided trigger and substrate ablation — RF based WACA ± electrophysiological testing guided ablation of non-PV triggers of AF and low voltage area ablation
  Arms: RF based WACA ± EP testing guided ablation of non-PV triggers of AF and low voltage area ablation

SUMMARY:
Atrial Fibrillation (AF) is a heart rhythm disturbance that affects over a million people in North America. AF can cause strokes, heart failure, poor quality of life and may lead to premature death. Catheter ablation has been shown to be superior to medications for symptoms, prevention of stroke and heart failure. AF recurrence is a problem after catheter ablation. Our research has found that in most cases AF recurrence occurs because the catheter procedure was ineffective. The objective of our clinical trial is to find out if a new method of performing the catheter procedure will be more effective in preventing AF recurrence compared to the current standard of care ablation procedure. Subjects will be randomly allocated to undergo either the standard of care ablation, or the novel patient tailored ablation. The novel method aims to understand the unique factors responsible for AF in each individual and uses this information to perform a patient-tailored catheter ablation procedure. This is expected to improve the results of AF ablation. The effectiveness and safety of the ablation procedure will be specifically evaluated in women to understand the effect of sex on AF ablation.

DETAILED DESCRIPTION:
Catheter ablation (CA) for paroxysmal atrial fibrillation (AF) is beset by the significant limitation of recurrent AF in one third of subjects. Subjects with recurrence of AF usually require repeat ablation procedures with the attendant risk of potentially serious complications and significant costs to the health care system. We hypothesize that an innovative, a patient specific precise CA strategy will significantly reduce AF recurrence.

This study will determine whether a precise, patient specific ablation strategy (tailored to the patient's triggers and substrate) combining electrophysiological (EPS) testing guided radiofrequency catheter ablation (RFA) for pulmonary vein isolation (PVI) using the wide-area circumferential (WACA) technique along with non-pulmonary vein trigger (NPVT) and low-voltage area (LVA) ablation will improve freedom from recurrent atrial fibrillation (AF) when compared to PVI alone strategy using cryoballoon ablation (CAB).

The PVI-WACA technique has a 'ceiling effect' due to PV reconnection, especially along the posterior wall of the LA as shown in an observational study investigating the pattern of PV reconnection from our institution. Further attempts at improving durable PVI rates with higher energy ablation may not be possible due to concerns regarding esophageal injury and development of atrio-esophageal fistula. It may be possible to improve the results of CA for paroxysmal AF by targeting NPVT and LVA that are not usually targeted during CA using the PVI-WACA only strategy.

This trial is a single-blinded (subjects blinded), prospective, parallel arm RCT. Subjects satisfying the inclusion and exclusion criteria will be randomized (1:1) to either the control arm (cryoballoon ablation) or the experimental arm (RF based WACA ± electrophysiological testing guided ablation of non-PV triggers of AF and low voltage area ablation). Randomization will be conducted after informed consent has been obtained and before catheter ablation. The first 60 days after catheter ablation will be considered a "blanking-period" and atrial tachyarrhythmias (AF, Atrial Flutter [AFl] or Atrial Tachycardia [AT]) occurring during this period will be documented. However, these will not be considered treatment failures. Subject accrual will occur over a 36-month period and each subject will have a minimum follow-up period of 24 months, with a total trial duration of 60-months. Subjects will be followed up at 2,6,12,18 and 24 months after ablation, with an implantable loop recorder (ILR) interrogation. Quality of life questionnaires (EQ-5D, AFEQT questionnaires and CCS-SAF scale) will be administered at baseline,12-months and 24 months post ablation visit. A tool to assist in decision making will be administered to subjects during the consent process.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years on the date of consent for the trial.
2. Subjects must have Paroxysmal AF with at least two episodes of AF over the past 12 months; Early Persistent AF- at least two episodes of AF.
3. At least one episode of AF documented on 12-lead ECG, Holter monitor, Trans- telephonic monitor (TTM) or Loop Recorder.
4. Subjects must be able to provide informed consent.

Exclusion Criteria:

1. Persistent and permanent AF
2. History of previous catheter or surgical ablation for AF, AFl, AT, AVNRT, AVRT.
3. Documented AVNRT, AVRT, AT or Atrial Flutter prior to enrolment in the trial.
4. Previous left atrial (LA) ablation or LA surgery.
5. Previous pulmonary vein stenosis or pulmonary vein stent.
6. Pre-existing hemi-diaphragmatic paralysis.
7. Active intracardiac thrombus.
8. Contraindication to systemic oral anticoagulation therapy or radiocontrast materials.
9. Current immunosuppressant therapy (corticosteroids, biologic immunomodulators; such patients may be considered if they can safely discontinue immunosuppressants for three months prior to and for three months following catheter ablation).
10. Reversible causes of AF (eg. uncontrolled hyperthyroidism, within six months of cardiac surgery).
11. Left ventricular ejection fraction <35%.
12. NYHA Class 3-4 heart failure.
13. Hypertrophic cardiomyopathy with septal or posterior LV wall thickness of >1.8 cm.
14. Significant valve disease (moderate or severe mitral/aortic stenosis or regurgitation).
15. Known adverse reaction to adenosine.
16. Significant chronic kidney disease (eGFR <30ml/min/1.73m2).
17. Significant congenital heart disease (including atrial septal defects or pulmonary vein abnormalities; however, subjects with patent foramen ovale will not be excluded).
18. Pregnant subjects.
19. Cerebral ischemic event (stroke or transient ischemic attack) in the six months prior to consenting for the trial.
20. Life expectancy less than one-year.
21. Currently participating or anticipated to participate in clinical trials of drug, device or biologic agents that could affect the results of this trial.
22. Unwilling or unable to comply fully with study procedures and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation, atrial flutter or atrial tachycardia | 61 to 365 days after ablation
  AF, AFl or AT, symptomatic or asymptomatic lasting ≥ 30 seconds

SECONDARY OUTCOMES:
Atrial fibrillation burden | 760 days
  Total duration of AF recorded on ambulatory monitoring/total duration of monitoring
Long-term rate of documented AF, AFl or AT | 760 days
  Long-term rate of documented AF, AFl or AT lasting ≥ 30 seconds
Incidence of any ECG/ILR documented AF, AFl or AT | First 60 days after catheter ablation
  Incidence of any ECG/ILR documented AF, AFl or AT (symptomatic or asymptomatic; lasting ≥ 30 seconds
Ablation procedure duration | On day of ablation
  Catheter ablation procedure time
Fluoroscopic exposure | On day of ablation
  Total Air Kerma (mGy)
Fluoroscopic exposure dose | On day of ablation
  Dose Area Protocol (Gy.cm2)
Procedure Related Complications | 760 days
  Stroke, PV stenosis, pericarditis, phrenic nerve palsy, cardiac perforation, atrio-esophageal fistula, major bleeding and/or death.
Emergency room visits or hospitalization due to recurrent AF, AFl or AT | 760 days
  Emergency room visits or hospitalization due to recurrent AF, AFl or AT
Repeat catheter ablation for AF, AFl or AT | 760 days
  Repeat catheter ablation for AF, AFl or AT
Quality of life scale | 12 and 24 months
  EQ-5D
Quality of life questionnaire | 12 and 24 months
  AFEQT questionnaire
Quality of life SAF scale | 12 and 24 months
  CCS-SAF scale

CONTACTS AND LOCATIONS:
Overall Officials: Girish Nair, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (2):
- Canada (2):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - McGill University Health Center, Montreal, Quebec